CLINICAL TRIAL: NCT00214617
Title: Effect of Crestor on the Kinetics of Plasma Apolipoproteins: Dose-Response Study
Brief Title: Effect of Crestor on Lipoprotein Metabolism in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Atlanta Veterans Education and Research, Inc. (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AREF_Le_IRUSROSU 0021; IRUSROSU 0021
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2006-09

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; HMG CoA Reductase Inhibtors; tracer kinetics; Apolipoproteins
MeSH Terms: conditions — Hypercholesterolemia

INTERVENTIONS:
Drug: Rosuvastatin at 5 mg/day and 40 mg/day

SUMMARY:
The objective of this research is to understand how Crestor can effectively reduce the levels of the bad cholesterol, LDL, in blood. It is hypothesized that with a low dose, Crestor will facilitate the rate of removal of LDL from the blood. At the higher dose, the increased potency of Crestor is explained by a reduction in the production of LDL by the liver.

DETAILED DESCRIPTION:
Crestor has been demonstrated to be effective in reducing plasma LDL by 20 to 60% in a dose dependent fashion. While the primary mechanism of action of this class of agents is the increase in the expression of LDL receptor resulting in accelerated clearance of LDL, the increase potency of Crestor in comparison to other statins may suggest other mechanisms. We propose to study the rate of incorporation of deuterated labeled leucine into VLDL apoB and LDL apoB and to determine the effect of two doses of Crestor (5 mg/day and 40 mg/day) on the production and clearance of apoB. Participants will be admitted to the General Clinical Research Center on three occasions (4 days, 3 nights per admission) for these metabolic studies. This is an open-label study design to reflect usual care with the first admission taking place while the participant is not on any lipid-lowering therapy. The second admission will occur after a minimum of 6 weeks on the low dose (5mg/day). The dose will be increased to 40 mg/day at the time of discharge and the third admission will occur after a minimum of 6 weeks on the higher dose.

A secondary objective of this study is to examine the rate of production and clearance of apoA-I, the major protein in HDL, at the 2 doses of Crestor. In addition to a reduction in LDL, Crestor has also been reported to result in a characteristic dose-dependent increase in HDL. The mechanism of this increase is not understood.

ELIGIBILITY:
Inclusion Criteria:

* TG between 200 and 400 mg/dL
* LDLc between 160 and 250 mg/dL
* HDLc between 30 and 50 mg/dL for men and 40-65 mg/dL for women
* Lp(a) less than 30 mg/dL
* Age between 50 and 75 years

Exclusion Criteria:

* current lipid-lowering therapy,
* primary hypertriglyceridemia (TG>400 mg/dL),
* High HDL (HDL>70),
* high Lp(a), greater than 30 mg/dL
* presence of beta-VLDL on agarose electrophoresis,
* current use of immunosuppressive agents,
* hormone replacement therapy for women
* history of cancer, active liver disease or hepatic dysfunction (AST or ALT 1.5 x ULN (Upper Limit of Normal),
* excessive consumption of alcohol, and recent history of drug abuse.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8
Dates: Start 2005-01; Study Completion 2006-02

PRIMARY OUTCOMES:
Rate of production of VLDL apoB
Rate of clearance of VLDL apoB
Rate of production of LDL apoB
Rate of clearance of LDL apoB

SECONDARY OUTCOMES:
Rate of production of HDL apoA-I
Rate of clearance of HDL apoA-I
Activity of cholesteryl ester transfer protein

CONTACTS AND LOCATIONS:
Overall Officials: Anh Le, PhD, Principal Investigator — Emory University School of Medicine and Atlanta VAMC
Locations (1):
- Atlanta Research and Education Foundation, Decatur, Georgia, United States